CLINICAL TRIAL: NCT01992718
Title: What Are we Missing? Diagnosing Uterine Adenomyosis Using Ultrasound Elastography
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Association of University Radiologists (Unknown); GE Radiology Research Academic Fellowship (Unknown)
Responsible Party: Principal Investigator, Katherine Maturen, M.D., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00076620
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Uterine Bleeding; Uterine Fibroids; Adenomyosis
MeSH Terms: conditions — Uterine Hemorrhage; Leiomyoma; Adenomyosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Evaluation of MRI, US for pelvic conditions (Active Comparator): MRI and ultrasound imaging will be used clinically to evaluate pelvic pain and abnormal uterine bleeding. The goal is to determine which exams are most helpful to the clinician in providing an accurate diagnosis as well as evaluating patient preference.
  Interventions: Procedure: Evaluation of MRI, US for pelvic and uterine conditions
- Patient preference MRI vs. US (Active Comparator): We are asking subjects to evaluate patient preference between MRI (magnetic resonance imaging) and ultrasound to determine which they would rather undergo.
  Interventions: Procedure: Patient preference between MRI and Ultrasound

INTERVENTIONS:
Procedure: Evaluation of MRI, US for pelvic and uterine conditions — Pelvic ultrasound with transabdominal and transvaginal imaging. The transvaginal ultrasound will include elastography (TVUS-E). Also, a pelvic MRI will be performed if not done in the last 6 months. The MRI is performed with IV gadolinium-based contrast (MultiHance ®).
  A patient survey will be included.
  Arms: Evaluation of MRI, US for pelvic conditions
Procedure: Patient preference between MRI and Ultrasound — Subjects may take part in this arm because they have recently had a MRI performed and scheduled for, or have recently undergone a pelvic ultrasound.
  Subjects will also be asked to complete a survey that will state their preference with regards to examination/imaging. This will be done over the phone and will take no longer than 30 minutes to complete.
  Arms: Patient preference MRI vs. US

SUMMARY:
To improve the clinical care of women with pelvic pain and abnormal uterine bleeding due to benign uterine conditions including leiomyomas (uterine fibroids) and adenomyosis by evaluating the accuracy of radiology diagnostic exams (MRI(magnetic resonance imaging), ultrasound and ultrasound with elastography).

DETAILED DESCRIPTION:
Currently benign conditions of the uterus are frequently underdiagnosed or misdiagnosed. This project will help determine which diagnostic radiology exams are most helpful to the clinician in providing accurate diagnosis. In addition, this study will evaluate which exam (MRI vs. Ultrasound) patients prefer over another exam.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Pelvic pain and/or abnormal uterine bleeding. (this is specific for Arm. 1 of this study)
3. If you have had or are scheduled to have both a pelvic MRI (magnetic resonance imaging) and a pelvic ultrasound with 6 months of the time of enrollment. (this is specific to Arm 2 of this study).

   -

Exclusion Criteria:

1. If you are post-menopausal(have not had a period in at least one year's time).
2. If you have been diagnosed with gynecological malignancy such as uterine, endometrial, cervical or ovarian cancer.
3. If you are unable or unwilling to sign the informed consents
4. If you are unable to undergo the research study exams -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of MRI and ultrasound elastography for distinguishing adenomyosis and fibroids | 1-2 months per patient
  Arm 1 patients will undergo hysterectomy (per previously defined clinical decision unrelated to the study) 4-6 weeks after enrollment and imaging tests, allowing us to correlate imaging and pathologic findings

SECONDARY OUTCOMES:
Patient preference between ultrasound and MRI | 6 months per patient
  Patients will take a survey to assess their experiences and preferences for pelvic imaging tests within 6 months after having those tests

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Maturen, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No